CLINICAL TRIAL: NCT06283160
Title: Interest of Metabolomic and Immune Profiling in the Development of Pancreatic Fistulas After Duodenopancreatectomy
Brief Title: METabolomic and Immune PROfiling in the Development of Pancreatic Fistulas After cepHalic duodEnopancreatectomy
Acronym: PROMETHEE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/834
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Fistula; Acute Pancreatitis; Pancreatoduodenectomy
Keywords: Metabolomics; Immune response; Pancreatic fistula; pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula; Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non tumoral pancreas (<0.2g) Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatoduodenectomy is the standard surgical operation for benign or malign pancreatic lesions. Pancreatic Fistula (PF) or Postpancreatectomy Acute Pancreatitis (PPAP) are the major complications associated with that type of surgery. We need to develop preventive measures for these complications, which requires a better understanding of their physiopathology.

The aim of this prospective monocentric and observational study is to identify predictive biomarkers and/or risk factors for PF or PPAP using metabolomics. The Profiling of circulating metabolites is indeed an original and promising approach for this purpose. We will also investigate the patient's immune status and its association with the occurrence of post-surgical complications.

Participants will be adult patients scheduled to undergo elective pancreaticoduodenectomy. Surgery and patient's management will be as usual. During surgery, a fragment (0.1-0.2 g) of non-tumoral pancreatic tissue will be removed and frozen at -80°C for metabolomic analysis. For immunological assessment, 4 blood samples will be collected (before surgery and then 7 days, 1 and 3 months after, blood sampling).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo elective pancreaticoduodenectomy
* Non-opposition of the subject to participate in the study.
* Affiliated to the French social security system (CMU included).

Exclusion Criteria:

* Emergent surgery.
* Pregnant patients.
* Refusal to participate or inability to provide informed consent.
* Patient under legal protection (individuals under guardianship by court order).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be made of adult patients scheduled to undergo elective pancreaticoduodenectomy in the University hospital of Besançon (France)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
occurrence of clinically significant FP and/or PAPP during hospitalization following pancreaticoduodenectomy. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Besançon, Besançon, France